CLINICAL TRIAL: NCT01331785
Title: Mechanism and the Effect of Midodrine on Portal Pressures in Patients With Cirrhosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: The Cleveland Clinic (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACG-CR-026-2010
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2011-04

CONDITIONS: Cirrhosis; End Stage Liver Disease; Ascites; Hypotension
Keywords: paracentesis; ascites; hypotension
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease; Ascites; Hypotension | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midodrine (Experimental)
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — Midodrine 2.5 mg to 10 mg three times a day to increase systolic BP above 100 mmHgor by 10 mmHg

SUMMARY:
Ascites is a frequent complication of patients with portal hypertension. As portal hypertension progresses, a percentage of these patients develop refractory ascites. Management options at that point include either TIPS or intermittent large volume paracentesis (LVP), with its attendant risks, Portal hypertension is accompanied by systemic circulatory dysfunction (decreased systemic vascular resistance and systolic BP), which is exacerbated by large volume paracentesis, with resultant renal and cardiac dysfunction. There are limited options for managing patients with acute decompensation, such as hepatorenal syndrome, although midodrine and other vasoconstrictors have been used in such patients. Midodrine has not been used as a possible therapeutic for ascites. Midodrine however, has been found to change the hemodynamics related to portal hypertension and ascites. There has been also change in mediators related to renal and circulation in studies of short duration (7 days) but not found in studies of 1 month duration, however the clinical effects of midodrine is found for longer duration in other similar conditions.

The purpose of the study is to assess the utility of midodrine in patients with obvious systemic circulatory dysfunction (hypotension) in improving the outcome of patients with refractory ascites and change in hemodynamic parameters and its mediators.

Specific endpoints include:

1) an objective reduction of the volume/rate of accumulation of ascites and 2) a decrease in the frequency of LVP.

DETAILED DESCRIPTION:
The pathophysiology of ascites is complex and various mechanisms have been proposed. Splanchnic and systemic vasodilation related to excess nitric oxide has been associated with systemic hypotension and increased portal flow.(8-10) This is associated with hemodynamic compensatory mechanisms, including activation of the renin-angiotension aldosterone system (RAAS), sympathetic nervous system (SNS), and non osmotic release of anti-diuretic hormones (ADH).(11, 12) These ultimately result in renal dysfunction, associated with sodium and fluid retention.(13) Several studies have shown reversal of HRS and decreased circulatory dysfunction when vasoconstrictors are administered. Various vasoconstrictors (noradrenaline, teleperessin, octreotide and midodrine) have been used in the management of hepato renal syndrome (HRS). (14-17) Midodrine appears to have some advantages, including the benefit of being an oral medication. (18) The beneficial effects have been noted as early as 6 hours after the use of midodrine in patients with ascites with or without HRS (2) with decreased plasma renin activity (PRA), antidiuretic hormone (ADH), nitrite and nitrate activity (NOx), increased renal plasma flow (RPF), glomerular filtration rate (GFR), increased urine sodium concentration (UNa) and volume, increased mean atrial pressure (MAP), decreased heart rate (HR) and cardiac output (CO). There was also decreased aldosterone in non-azotemic cirrhotic patients with or without ascites in patients studied for 7 days. (3) The renal function improvement was not substantiated in other studies. In patients treated for a month along with octreotide there was no significant improvement of renal function but marginal reversible liver dysfunction with decreased body weight (paracentesis adjusted weight),(19) A similar significant weight reduction was also noted in another study.(7) Midodrine has been shown to be safe and effective in patients when used to prevent dialysis induced hypotension, and has improved systolic pressure, without a significantly increased volume of fluid filtered by dialysis and no change in body weight in patients studied.(20, 21) The beneficial effects have been attributed to its modulating effects on autonomic function and increasing peripheral vessel resistances.(22) The drug has been found to effective and safe in acute and chronic use (21, 23) with minimal side effects.(24)

Vasoconstrictors in patients with ascites and hydrothorax In non azotemic cirrhotic patients with ascites, the addition of octreotide improved diuresis and decreased renin, increased MAP, decreased CO and improved renal function by increasing GFR, increased urine sodium and volume excretion.(25) In patient with massive hydrothorax with mild ascites and no azotemia, addition of midodrine to octreotide improves MAP, increases GFR, RPF and urine sodium and volume; and prevents recurrence of hydrothorax. Vasoconstrictors have been recommended as treatment for hydrothorax (4-6)and has been found beneficial in refractory ascites.(26)

Significance Vasoconstrictors like midodrine have been shown to be beneficial, with improvement of circulatory dysfunction in various groups of patients including patients with HRS type 1, type 2, non azotemic patients and in patients requiring hemodialysis. There are suggestions of decreased body weight in some of these patients. In patients with hydrothorax, addition of vasoconstrictors has helped in relieving the symptoms. The investigators suggest that midodrine could also benefit patients with refractory ascites. By decreasing the rate of ascitic fluid accumulation, it may be possible to decrease the volume of ascites drained or lengthen the interval between paracentesis, giving comfort to the patients. The beneficial effect on portal pressures and ascites could be due to other mechanisms (such as autonomic function) rather than their effect on renal hemodynamics as they are not sustained. There are no studies where this has been systematically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old
* Evidence of ESLD and ascites
* Ascites requiring periodic large volume paracentesis (1+ / month) of more than 3 months duration
* Systolic BP < 100 mmHg

Exclusion Criteria:

* Prior liver transplant
* Evaluated for multiple organ transplant
* Malignancies
* Non cirrhotic causes of ascites
* Prior TIPS usage (transjugular intrahepatic porto-systemic shunt)
* Primary renal diseases
* Chronic kidney disease (CKD) >=4
* Grade 3 or 4 encephalopathy
* Child C cirrhosis or model for end stage liver disease (MELD) > 20
* Patients requiring large volume paracentesis for more than 12 months
* Frequency of paracentesis less than 6 in the preceding 3 months
* Active recreational drug and alcohol usage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Volume and frequency of paracentesis and quality of life | 3 months of study drug
  To quantify the volume and rate of production of ascites (as estimated by the frequency of paracentesis) in patients with refractory ascites and hypotension requiring intermittent LVP and comparing these values before and after use of midodrine.

SECONDARY OUTCOMES:
Renal and cardiovascular hemodynamic changes | 3 months
  2. To determine the effect of midodrine on the hemodynamics in these patients as well us its effect on circulatory (blood pressure), renal parameters (BUN, creatinine, serum and urine sodium), and the hormones and mediators (plasma renin, anti diuretic hormone, angiotension, aldosterone, nitrite and nitrate activity) known to be associated with cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Achuthan Sourianarayanane, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States